CLINICAL TRIAL: NCT05586919
Title: Treatment of Venous Malformation by Direct Puncture Repair: Ethanol Versus Polidocanol
Brief Title: Treatment of Venous Malformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Walied Khereba, Principal Investigator, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Venous Malformation
Record Dates: First submitted 2022-10-01; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Venous Malformation
MeSH Terms: interventions — Ethanol; Polidocanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Puncture Repair / Ethanol (Active Comparator)
  Interventions: Procedure: Direct Puncture Repair / Ethanol
- Direct Puncture Repair / Polidocanol (Active Comparator)
  Interventions: Procedure: Direct Puncture Repair / Polidocanol

INTERVENTIONS:
Procedure: Direct Puncture Repair / Ethanol — Ethanol is an organic compound that will be injected in the venous malformation as a sclerotherapy by Direct Puncture Repair
  Arms: Direct Puncture Repair / Ethanol
Procedure: Direct Puncture Repair / Polidocanol — Polidocanol is a sclerosing agent that will be injected in the venous malformation by Direct Puncture Repair
  Arms: Direct Puncture Repair / Polidocanol

SUMMARY:
Vascular malformations are birth defects that happen when different stages of angiogenesis shut down. 44 - 64% of all vascular malformations are venous malformations (VMs). Sclerotherapy is the first treatment line for VMs. It acts by getting rid of the vascular endothelial cells in the lesion. One of the most common and well researched sclerosing agents for VMs is polidocanol, which is a popular counterpart for concentrated ethanol.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with venous malformation of both genders and age above one year.

Exclusion Criteria:

* Age below one year.
* Patients had any other vascular malformations.
* Indication for contrast material or Alcohol and polidocanol injection.
* Unfit for general anesthesia. 5) Pregnancy. 6) Skin infection, inflammation, and ulcers.
* Pulmonary embolism.
* Acute Ischemia, and acute DVT.

Ages: 18 Months to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Heaviness questionnaire | 6 months post operative
  Heaviness of the affected part may be unchanged, or decreased or disppeared, or relapsed
Disfigurement questionnaire | 6 months post operative
  Disfigurementof the affected part may be unchanged, or decreased or disppeared, or relapsed
size of venous malformation | 6 months post operative
  it assess the size of malformations after injection; which may be unchanged, or decreased or disppeared, or relapsed
Degree of satisfaction | 6 months post operative
  It may be; Very satisfied, or satisfied, or not satisfied, or Dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Walied Khereba, Zagazig, Egypt